CLINICAL TRIAL: NCT00326638
Title: Randomized Phase III Trial of 3D Conformal Radiotherapy Versus Helical Tomotherapy IMRT in High-Risk Prostate Cancer
Brief Title: 3D-Conformal Radiation vs Helical Tomotherapy in Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005242-01H; OTT 05-02
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: prostate, IMRT, tomotherapy, radiation, cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: 3D-Conformal Radiation (Other): Intervention: Standard radiation treatment for high risk prostate cancer. Once daily Monday to Friday for 8 weeks.
  3DCRT 7800 cGY/39 Fractions/ STD Technique*
  * Initial 4F 3DCRT to Nodes/ Prostate + Seminal Vesicles 4,600 cGy/23
  * Boost 6 F 3DCRT to Prostate 3,200 cGy/16
  Interventions: Other: Arm A: 3D-Conformal Radiation
- Arm B: Helical Tomotherapy Intensity Modulated Radiotherapy (Experimental): Intervention: Helical Tomotherapy Intensity Modulated Radiotherapy (IMRT) once daily Monday to Friday for 8 weeks.
  IMRT using Helical Tomotherapy* 7800 cGY/39 Fractions Boost IMRT to Prostate 3,200 cGy/16
  Interventions: Radiation: Arm B: Helical Tomotherapy Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Arm B: Helical Tomotherapy Intensity Modulated Radiotherapy — IMRT using Helical Tomotherapy* 7800 cGY/39 Fractions once daily Monday to Friday for 8 weeks
  * Initial IMRT to Nodes/Prostate + Seminal Vesicles 4,600 cGy/23
  * Boost IMRT to Prostate 3,200 cGy/16
  Other Names: IMRT
  Arms: Arm B: Helical Tomotherapy Intensity Modulated Radiotherapy
Other: Arm A: 3D-Conformal Radiation — 3DCRT 7800 cGY/39 Fractions/ STD Technique* once daily Monday to Friday for 8 weeks
  * Initial 4F 3DCRT to Nodes/ Prostate + Seminal Vesicles 4,600 cGy/23
  * Boost 6 F 3DCRT to Prostate 3,200 cGy/16
  Other Names: Radiation Therapy
  Arms: Arm A: 3D-Conformal Radiation

SUMMARY:
In this study we are comparing two forms of radiotherapy. This study is being done because it is not clear at present time whether intensity modulated radiotherapy (IMRT) can reduce side effects of radiotherapy compared to standard radiotherapy (called 3D-Conformal Radiotherapy).

DETAILED DESCRIPTION:
Radical radiation therapy plays an important role in the management of prostate cancer, yielding comparable long-term outcomes to surgery. Unfortunately, long term disease free survival data using PSA criteria have shown that less than 50% of high-risk patients are free of disease at 10 years. To improve on the results of conventional dose radiotherapy dose escalation with three-dimensional conformal radiation has been employed. Due to the irregular shape of the prostate and the variable motion of this organ there is substantial radiation of adjacent normal surrounding tissue during treatment which results in radiation-induced toxicity. Intensity-modulated radiation therapy (IMRT) is a new form of radiation therapy. Preliminary evidence suggests that IMRT improves the dose distribution during radiation therapy of the prostate. The hypothesis of this study is that IMRT delivered using Helical Tomotherapy can reduce late toxicity of radical radiotherapy as compared to three-dimensional conformal radiation (3DCRT) in high-risk prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. A pathologic diagnosis of adenocarcinoma of the prostate
2. Age greater than 18 years
3. ECOG performance status of 2 or less.
4. Presence of any of the following high risk features:

   * Clinical stage cT3-4 or
   * Gleason score 8-10 or
   * Pre-treatment PSA > 20ng/ml or
   * Clinical N1/N2 or pathologic N1/N2

Exclusion Criteria:

1. Patients with contraindication to radical radiation therapy including inflammatory bowel disease
2. Prior or active malignancy except non-melanoma skin carcinoma within 5 years of the diagnosis of prostate cancer
3. Prior pelvic radiotherapy for other malignancies
4. Prior cytotoxic chemotherapy
5. Prior orchiectomy, radical prostatectomy, cryotherapy or thermal ablation therapy for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2005-03; Primary Completion 2015-01 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Late rectal toxicity from radiotherapy of the prostate | Month 1, 4, 8, every 4 months during year 1-2, then every 6 months during years 2-5, then every 12 months until disease progression
  Outcome measurements will be determined by physical exam and bloodwork.

SECONDARY OUTCOMES:
Acute rectal toxicity, Acute and late bladder toxicity, Disease specific survival at 5 years, Biochemical relapse free survival at 5 years, Local control rates at 5 years, Quality of Life | Month 1, 4, 8, every 4 months during year 1-2, then every 6 months during years 2-5, then every 12 months until disease progression
  Outcome measurements will be determined by physical exam and bloodwork.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Malone, MD, Study Director — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario, Canada